CLINICAL TRIAL: NCT00787995
Title: A Multicenter, Multinational, Longitudinal Clinical Assessment Study of Subjects With Mucopolysaccharidosis IVA (Morquio Syndrome)
Brief Title: A Clinical Assessment Study of Subjects With Mucopolysaccharidosis IVA (Morquio Syndrome)
Status: Terminated | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: MOR-001
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: MPS IV A; Mucopolysaccharidosis IVA; Morquio A Syndrome
Keywords: Mucopolysaccharidosis IV type A; MPS IV Type A; Mucopolysaccharidosis IVA; MPS IVA; Morquio A Syndrome; Lysosomal Storage Disorder; LSD; N-acetylgalactosamine-6-sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT
MeSH Terms: conditions — Mucopolysaccharidosis IV; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MPS IVA: Subjects with mucopolysaccharidosis IVA (Morquio Syndrome)

SUMMARY:
This multicenter, multinational, longitudinal study will quantify endurance and respiratory function in subjects diagnosed with MPS IVA and will better characterize the spectrum of symptoms and biochemical abnormalities in MPS IVA disease over time.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent, or in the case of subjects age < 18 years, provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
* Documented history of reduced GALNS activity relative to the normal range of the laboratory performing the assay, or documented result of molecular genetic testing confirming diagnosis of MPS IVA.
* Willing and able to comply with all study procedures.

Exclusion Criteria:

* Use of any investigational product or investigational medical device within 30 days prior to screening.
* Previous hematopoietic stem cell transplant (HSCT).
* Concurrent disease or condition that would interfere with study participation or pose a safety concern.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects diagnosed with MPS IVA
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2008-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Endurance | Study Visit
Respiratory Function | Study Visit

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Decker, MD, Study Director — BioMarin Pharmaceutical
Locations (15):
- United States (2):
  - Oakland, California
  - Chicago, Illinois
- Córdoba, Argentina
- Brazil (2):
  - Porto Alegre
  - São Paulo
- Montreal, Quebec, Canada
- France (2):
  - Lyon
  - Paris
- Mainz, Germany
- Monza, Italy
- Amsterdam, Netherlands
- Taipei, Taiwan
- United Kingdom (3):
  - Birmingham
  - London
  - Manchester

REFERENCES:
- [Derived] Martell LA, Cunico RL, Ohh J, Fulkerson W, Furneaux R, Foehr ED. Validation of an LC-MS/MS assay for detecting relevant disaccharides from keratan sulfate as a biomarker for Morquio A syndrome. Bioanalysis. 2011 Aug;3(16):1855-66. doi: 10.4155/bio.11.172. PMID 21877895
- See also: BioMarin Pharmaceutical Inc. website — http://www.bmrn.com